CLINICAL TRIAL: NCT02347826
Title: Evaluation of Aesthetic Satisfaction in Patients Undergoing Non Surgical Face and Neck Lift by Means of Coned Wires.
Brief Title: Evaluation of Satisfaction in Patients Undergoing Non Surgical Lifting by Means of Coned Wires.
Acronym: SCW
Status: Completed | Type: Observational
Sponsor: AQ-DE (Other)
Responsible Party: Sponsor
Other Study IDs: Aqde
Record Dates: First submitted 2015-01-21; First posted 2015-01-27 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Pain; Complications
Keywords: coned wires, wire lift,; patient; discomfort
MeSH Terms: conditions — Pain

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
An email questionnaire about subjective satisfaction and discomfort has been sent to 243 patients undergoing non-surgical facial and cervical lift 1 week, 1 month, 6 months and 1 year after treatment.

DETAILED DESCRIPTION:
243 patients underwent non-surgical coned wires (silhouette soft) facial and cervical lift between October 2013 and November 2014. The procedures has been executed in our aesthetic clinics in Milan, Bologna, Turin, Genoa, Rome, Asti, San Remo and Palermo.

Among the 243 patients, 217 were females and 26 males, with age ranging from 19 to 76 years. 103 patients underwent only facial lift, of which 12 only in the frontal area, 61 only on cheek and malar area, and 30 on both the areas.

39 patients underwent only cervical lift, of those 14 by means of appliance of 1 or 2 wires, 25 by means of appliance of more than 2 wires.

101 patients underwent both facial and cervical non surgical lift. We sent to every patient a email questionnaire1 week, 1 month, 6 months and 1 year after treatment.

In the questionnaire, patients has been asked to enter a value between 1 and 5 about subjective satisfaction regarding the aesthetic improvement (ranging from 1, poor, to 5, excellent), and discomfort related to treatment (ranging from 1, no perceived discomfort, to 5, impossibility to execute working and social activities).

The data has been analyzed and related to other factors such as:

* number of wires applied on each patient
* other aesthetic or regenerative medicine treatments executed on the same patient on the same year
* total expenditure related to aesthetic treatments in the same year

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing facial and cervical non surgical lift by means of resorbable coned wires

Exclusion Criteria:

* Patients with asymmetry

Ages: 19 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing non surgical facial and carvical lift from 2013 to 2014
Sampling Method: Non-Probability Sample
Enrollment: 243 (Actual)
Dates: Start 2014-01; Primary Completion 2014-01 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Subjective satisfaction questionnaire | up to one year

SECONDARY OUTCOMES:
Discomfort related to treatment questionnaire | one week, one month, 6 months, one year

CONTACTS AND LOCATIONS:
Overall Officials: Mario Goisis, MS, Study Director — AQ-DE
Locations (1):
- AQCE, Milan, Lombardia\Milan, Italy